CLINICAL TRIAL: NCT06208618
Title: The Effect of Education and Motivational Interviews Conducted Through Tele-Nursing on Diabetes Management in Adolescents With Type 1 Diabetes: A Randomized Controlled Trial
Brief Title: The Impact of Motivational Interviews Conducted Through Tele-Nursing on Diabetes Management
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Pınar Duru, Associate Professor, Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: YesimKorkusuz
Record Dates: First submitted 2024-01-06; First posted 2024-01-17 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Type 1 Diabetes; Motivational Interviewing
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: A single-center, single-blind, parallel-group, randomized controlled design
Who Masked: Participant
Masking Description: Single-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational interviews (Experimental): At the beginning of the study, individual face-to-face diabetes education will be provided for each adolescent in the study group on days corresponding to their routine medical appointments in the diabetes education room. The diabetes education will include the following topics:
  * What is Diabetes?
  * Treatment in Diabetes
  * Insulin Therapy
  * Nutritional Therapy
  * Physical Activity/Exercise
  * Acute Complications of Diabetes
    * Hypoglycemia
    * Hyperglycemia
    * Diabetic Ketoacidosis
  * Diabetes Management in IIlness
  The adolescents in the study group will undergo a total of 6 motivational interviews, conducted once a month. Three of these interviews will be face-to-face (at the beginning of the study, at the 3rd month, and at the 6th month), while the remaining three will be conducted remotely using the WhatsApp video call feature (in the 2nd, 4th, and 5th months).
  Interventions: Other: Education and Motivational Interviews
- Routine follow-up (No Intervention): The routine follow-up conducted by the diabetes education unit will continue for the study group, and no interventions will be made as part of the research. The study group will undergo a pre-test at the beginning of the study, a follow-up test at the 3rd month, and a post-test at the 6th month as part of the research.

INTERVENTIONS:
Other: Education and Motivational Interviews — The diabetes education aimed at supporting diabetes self-management in adolescents will include the following topics:
  * What is Diabetes?
  * Treatment in Diabetes
  * Insulin Therapy
  * Nutritional Therapy
  * Physical Activity/Exercise
  * Acute Complications of Diabetes
    * Hypoglycemia
    * Hyperglycemia
    * Diabetic Ketoacidosis
  * Diabetes Management in Illness
  Motivational interviews will consist of the following stages:
  * First Meeting - Pre-awareness (Pre-contemplation)
  * Second Meeting - Awareness (Contemplation)
  * Third Meeting - Preparation
  * Fourth Meeting - Taking Action (Action)
  * Fifth Meeting - Maintenance
  * Sixth Meeting - Termination or Review
  Arms: Motivational interviews

SUMMARY:
The deterioration of glycemic control in adolescents with Type 1 diabetes (T1DM) is a genuine cause for concern. Possible reasons for worsening glycemic control in youth include lack of monitoring, inadequate self-care, psychosocial factors, lack of family support and parental supervision, non-adherence to treatment, pubertal increases in insulin resistance, and insufficient transition from pediatric to adult care. In adolescents with established T1DM who transition to adult-focused care, there is observed disengagement or complete detachment from care. Improving glycemic control during adolescence is a critical stage to enhance and reduce complications associated with T1DM. Adolescents with T1DM require appropriate daily insulin therapy, regular blood sugar monitoring, physical activity, healthy nutrition, education, and support to delay or prevent diabetes-related complications.This study aims to determine the impact of education and motivational interviews conducted through tele-nursing on the management of diabetes in adolescents with Type 1 diabetes.

DETAILED DESCRIPTION:
The study will be conducted with a single-center, single-blind, parallel-group, randomized controlled design with a follow-up period of 6 months.The population of the study consists of 141 adolescents aged 13-18 diagnosed with Type 1 diabetes, who are being followed up at the Diabetes Education Unit of Evliya Çelebi Training and Research Hospital, affiliated with Kütahya Health Sciences University in the province of Kütahya, Türkiye. The sample of the study will consist of 96 adolescents, with 48 participants in each group, assuming a 1:1 randomization, based on the reference study. In their research, where motivational interviews were used for adolescents' diabetes management, the reported HbA1c levels for the study group (9.61±2.40) and the control group with routine follow-up (10.76±2.07) at the 6-month follow-up were considered, aiming for an 80% power and a 0.05 margin of error.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Type 1 diabetes at least 6 months ago
* Under follow-up at Kütahya Evliya Çelebi Health Sciences University Training and Research Hospital Diabetes Education Unit
* Having an HbA1c level above 7.5% in the most recent measurement
* Having a smartphone

Exclusion Criteria:

* Refusal of legal guardian or the adolescent themselves to participate in the research
* Difficulty in communication or answering questions
* Having hearing, speech, vision, or cognitive impairments
* Being in the honeymoon period of Type 1 diabetes
* Having a second autoimmune disease, such as celiac disease, besides Type 1 diabetes

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
HbA1c level | At the beginning of the study, at the 3rd month, and at the 6th month
  HbA1c level
Diabetes management self-efficacy | At the beginning of the study, at the 3rd month, and at the 6th month
  It will be measured using the "Diabetes Management Self-Efficacy Scale in Adolescents with Type 1 Diabetes". The scale consists of a total of 26 items under four sub-dimensions named "medical treatment and nutrition", "glycemic assessment", "talking about your diabetes" and "honesty towards yourself and others".The items in the scale are answered according to the 5-point Likert system as "Definitely yes (1) - Definitely no (5)". Self-efficacy scores are summed and divided by the total number of items to indicate the strength of perceived self-efficacy for different levels of performance on the total of diabetes self-management activities. High scores on the scale represent low self-efficacy. The Cronbach Alpha reliability coefficient of the overall scale is 0.85; for the sub-dimensions are 0.80, 0.75, 0.70 and 0.70, respectively.

SECONDARY OUTCOMES:
Belief in a healthy lifestyle | At the beginning of the study, at the 3rd month, and at the 6th month
  It will be measured using the Healthy Lifestyle Belief Scale for Adolescents. The scale consists of a total of 16 items under three sub-dimensions named "health belief", "physical activity" and "nutrition". The items in the scale are answered according to the 5-point Likert system as "Strongly disagree (1) - Strongly agree (5)". A minimum of 16 and a maximum of 80 points can be obtained from the scale, and increasing scores from the scale indicates that adolescents' belief in a healthy life has increased. The Cronbach Alpha reliability coefficient of the overall scale is 0.90; for the sub-dimensions are 0.84, 0.79 and 0.81, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Pınar Duru, Ph.D., Principal Investigator — Eskisehir Osmangazi University
Locations (1):
- Eskisehir Osmangazi University, Eskişehir, Odunpazarı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No